CLINICAL TRIAL: NCT01255969
Title: EXerCise Introduction To Enhance Performance in Dialysis: the EXCITE Study
Brief Title: EXerCise Introduction To Enhance Performance in Dialysis(EXCITE)
Acronym: EXCITE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Principal Investigator, Carmine Zoccali, prof., Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXCITE-001
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Patients on Dialysis (Hemodialysis, Peritoneal Dialysis)
Keywords: Dialysis; Physical exercise; Clinical Trial; Quality of Life; Performance; Fitness; Cardiovascular Mortality; Vascular access
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- Exercise (Experimental): Patients in this arm will undergo to personalized exercise program.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Personalized exercise program
  Arms: Exercise

SUMMARY:
To evaluate if a model of intervention based on a low-grade physical program prescribed in the dialysis centre and performed at home can modify the functional capacity and quality of life, reduce the risk of cardiovascular and all-causes mortality, non-fatal cardiovascular events and vascular access failure in dialysis patients.

DETAILED DESCRIPTION:
Background Dialysis patients show an exceedingly higher risk of death and cardiovascular complications (1). These patients are also characterized by poor physical performance and reduced quality of life. Observational findings in the United States Renal Data System (USRDS) indicated that physical rehabilitation programs after coronary artery bypass are associated with better clinical outcomes in this population (2). However, the hypothesis that physical training in dialysis patients may translate into better physical performance and clinical outcomes has never been tested in large randomized clinical trials. In studies performed so far, physical exercise was proposed during the dialysis session or between two dialysis sessions. These programs imply compliance, organization and cost problems, mainly related with intensification of visit to the dialysis centre. To limit these difficulties, a single easy-to-implement program of physical exercise for dialysis patients, prescribed in the dialysis centre but performed at home, has been recently elaborated and a pilot study has shown that this program improves physical performance in medium term (3).

Purpose This clinical trial tests whether a physical program prescribed in the dialysis centre but performed at home improves the degree of fitness and the quality of life in dialysis patients.

Study population

* Inclusion Criteria:

  * 500 Patients on dialysis
  * Dialysis vintage>6 months
  * Age>18 years
  * Signed informed consent
  * Stable clinical conditions
* Exclusion Criteria:

  * physical or clinical limitations to deambulation

Outcomes:

* Functional capacity : Evaluation of the variation in the distance covered in a pre-determined time with a validated walking test (six minute walking test); Evaluation of the variation in the time needed to complete 5 cycles of the "sit-to-stand-to sit" test.
* Quality of Life : Score obtained by a validated questionnaire for dialysis patients (Kidney Disease Quality of Life instrument o KDQOL).
* Fatal and non-fatal events (cardiovascular and all-causes).
* All-cause hospitalizations.
* Vascular access survival. The power analysis was performed by calculating the sample size for each clinical outcome contemplated by the study protocol. The overall sample size of the trial is that portended by the calculation demanding the highest individuals numbers (that of the outcome "fatal and non fatal cardiovascular events" in our instance).

In a previous observational study by our group, the incident rate of fatal and non fatal cardiovascular events was at three years 25% (4). We hypothesised that the physical exercise will produce a 10% reduction in the hazard ratio of fatal cardiovascular events (hazard ratio: 0.70) as compared to that of the control group.

References:

1. Mallamaci F, Tripepi G, Cutrupi S, Malatino LS, Zoccali C. Prognostic value of combined use of biomarkers of inflammation, endothelial dysfunction, and myocardiopathy in patients with ESRD. Kidney Int. 2005 Jun;67(6):2330-7. PMID: 15882276
2. Kutner NG, Zhang R, Huang Y, Herzog CA. Cardiac rehabilitation and survival of dialysis patients after coronary bypass. J Am Soc Nephrol. 2006 Apr;17(4):1175-80. Epub 2006 Feb 15. PMID: 16481413
3. Malagoni AM, Catizone L, Mandini S, Soffritti S, Manfredini R, Boari B, Russo G, Basaglia N, Zamboni P, Manfredini F. Acute and long-term effects of an exercise program for dialysis patients prescribed in hospital and performed at home. J Nephrol. 2008 Nov-Dec;21(6):871-8. PMID: 19034871
4. Zoccali C, Tripepi G, Mallamaci F.Predictors of cardiovascular death in ESRD.Semin Nephrol. 2005 Nov;25(6):358-62

ELIGIBILITY:
Inclusion Criteria:

* Patients on dialysis
* Dialysis vintage>6 mo.
* Age>18 aa.
* Signed informed consent
* Stable clinical conditions

Exclusion Criteria:

-any physical or clinical limitations to deambulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-04; Primary Completion 2014-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Assessment of Quality of Life (QoL) modification by the KIDNEY DISEASE QUALITY OF LIFE (KDQOL)questionary | 6 months
  6 months is the time frame for the primary analysis but the follow-up will continue until 3 years.
Assessment of functional capacity by Six-Minute Walking test and Sit-to-Stand-to-sit test | 6 months
  6 months is the time frame for the primary analysis but the follow-up will continue until 3 years.

SECONDARY OUTCOMES:
Evaluation of mortality (all causes and cardiovascular only), non-fatal cardiovascular events, all-causes hospitalizations and dialysis access survival. | 6 months
  6 months is the time frame for the primary analysis but the follow-up will continue until 3 years.
All - causes and cardiovascular hospitalizations | 6 months
  Hospitalizations will be characterized by ICD-9 codes. Six months is the time frame for the primary analysis but the follow-up will continue until 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Zoccali, Prof., Study Director — CNR-IBIM and Nephrology Unit, Reggio Calabria
Locations (1):
- Dialysis Units participating to the EXCITE study in Italy, Reggio Calabria, Italy

REFERENCES:
- [Background] Mallamaci F, Tripepi G, Cutrupi S, Malatino LS, Zoccali C. Prognostic value of combined use of biomarkers of inflammation, endothelial dysfunction, and myocardiopathy in patients with ESRD. Kidney Int. 2005 Jun;67(6):2330-7. doi: 10.1111/j.1523-1755.2005.00338.x. PMID 15882276
- [Background] Kutner NG, Zhang R, Huang Y, Herzog CA. Cardiac rehabilitation and survival of dialysis patients after coronary bypass. J Am Soc Nephrol. 2006 Apr;17(4):1175-80. doi: 10.1681/ASN.2005101027. Epub 2006 Feb 15. PMID 16481413
- [Background] Malagoni AM, Catizone L, Mandini S, Soffritti S, Manfredini R, Boari B, Russo G, Basaglia N, Zamboni P, Manfredini F. Acute and long-term effects of an exercise program for dialysis patients prescribed in hospital and performed at home. J Nephrol. 2008 Nov-Dec;21(6):871-8. PMID 19034871
- [Derived] Mallamaci F, Bratsiakou A, D'Arrigo G, Tripepi G, Lamberti N, Torino C, Manfredini F, Zoccali C. Sex Differences in the EXerCise Introduction to Enhance Performance in Dialysis Trial. Clin J Am Soc Nephrol. 2025 Jun 13;20(8):1072-1078. doi: 10.2215/CJN.0000000759. PMID 40512565
- [Derived] Mallamaci F, D'Arrigo G, Tripepi G, Lamberti N, Torino C, Manfredini F, Zoccali C. Long-Term Effect of Physical Exercise on the Risk for Hospitalization and Death in Dialysis Patients: A Post-Trial Long-Term Observational Study. Clin J Am Soc Nephrol. 2022 Aug;17(8):1176-1182. doi: 10.2215/CJN.03160322. Epub 2022 Jul 25. PMID 35878932
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Baggetta R, D'Arrigo G, Torino C, ElHafeez SA, Manfredini F, Mallamaci F, Zoccali C, Tripepi G; EXCITE Working group. Effect of a home based, low intensity, physical exercise program in older adults dialysis patients: a secondary analysis of the EXCITE trial. BMC Geriatr. 2018 Oct 20;18(1):248. doi: 10.1186/s12877-018-0938-5. PMID 30342464
- [Derived] Manfredini F, Lamberti N, Malagoni AM, Felisatti M, Zuccala A, Torino C, Tripepi G, Catizone L, Mallamaci F, Zoccali C. The role of deconditioning in the end-stage renal disease myopathy: physical exercise improves altered resting muscle oxygen consumption. Am J Nephrol. 2015;41(4-5):329-36. doi: 10.1159/000431339. Epub 2015 Jun 11. PMID 26067552
- [Derived] Torino C, Manfredini F, Bolignano D, Aucella F, Baggetta R, Barilla A, Battaglia Y, Bertoli S, Bonanno G, Castellino P, Ciurlino D, Cupisti A, D'Arrigo G, De Paola L, Fabrizi F, Fatuzzo P, Fuiano G, Lombardi L, Lucisano G, Messa P, Rapana R, Rapisarda F, Rastelli S, Rocca-Rey L, Summaria C, Zuccala A, Tripepi G, Catizone L, Zoccali C, Mallamaci F; EXCITE Working Group. Physical performance and clinical outcomes in dialysis patients: a secondary analysis of the EXCITE trial. Kidney Blood Press Res. 2014;39(2-3):205-11. doi: 10.1159/000355798. Epub 2014 Jul 29. PMID 25118076